CLINICAL TRIAL: NCT00855686
Title: A Randomised, Double-blind, Placebo-controlled, 6-month Study of the Efficacy and Safety of Memantine in Patients With Parkinson's Disease Dementia or Dementia With Lewy Bodies
Brief Title: Memantine Versus Placebo in Parkinson's Disease Dementia or Dementia With Lewy Bodies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11018; 2005-002038-36 (EudraCT Number)
Record Dates: First submitted 2009-03-03; First posted 2009-03-04 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-09

CONDITIONS: Parkinson's Disease Dementia; Dementia With Lewy Bodies
Keywords: Memantine; Cognition; Parkinson's Disease Dementia; Dementia With Lewy Bodies
MeSH Terms: conditions — Lewy Body Disease | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Memantine (Experimental)
  Interventions: Drug: Memantine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Memantine — 20mg once daily oral dose
  Other Names: Ebixa®
  Arms: Memantine
Drug: Placebo — Daily oral dose
  Arms: Placebo

SUMMARY:
The purpose of this exploratory study is to determine whether memantine can provide benefits on clinical symptoms in patients with Parkinson's Disease Dementia or Dementia with Lewy Bodies.

DETAILED DESCRIPTION:
The objective of this exploratory study is to assess the benefits of memantine compared to placebo in out-patients with a diagnosis of Parkinson's Disease Dementia or Dementia with Lewy Bodies (mild to moderate severity) over a 6-month period. This is a multinational, randomised, double-blind, parallel-group, placebo-controlled, fixed-dose study with specific cognitive (attention, executive function, visual perception and memory), behavioural, functional and global measures.

ELIGIBILITY:
Inclusion Criteria:

* The study population will consist of male or female outpatients at least 50 years of age with mild to moderate disease severity (MMSE 12 to 24 inclusive) according to UKPDS and DSM IV TR criteria (for PDD patients) and the third report of the DLB consortium (for DLB patients) and who have a knowledgeable and reliable caregiver to accompany the patient to all clinic visits during the course of the study.

Exclusion Criteria:

* Evidence of clinically significant active disease, evidence of other neurological disorders, and current treatment with AChEIs.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2007-01; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
No primary or secondary outcome measures are defined. This study is exploratory (see above under detailed description).

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (1):
- DE001, Munich, Germany

REFERENCES:
- [Result] Emre M, Tsolaki M, Bonuccelli U, Destee A, Tolosa E, Kutzelnigg A, Ceballos-Baumann A, Zdravkovic S, Bladstrom A, Jones R; 11018 Study Investigators. Memantine for patients with Parkinson's disease dementia or dementia with Lewy bodies: a randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2010 Oct;9(10):969-77. doi: 10.1016/S1474-4422(10)70194-0. Epub 2010 Aug 20. PMID 20729148